CLINICAL TRIAL: NCT00505401
Title: A Phase I Safety and Immunogenicity Trial of Recombinant HIV-1 Tat in HIV-1 Infected Adult Volunteers
Brief Title: Phase I Safety and Immunogenicity Vaccine Trial Against HIV/AIDS
Acronym: ISST-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Responsible Party: Barbara Ensoli, MD, PHD, Istituto Superiore di Sanita
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISST-001
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2007-07

CONDITIONS: HIV Infections
Keywords: HIV; Tat protein; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Subjects were immunized subcutaneously with Tat, 3 dosage groups (7.5, 15 or 30 microgrammi), in association with Alum as adjuvant, or with Saline + Alum, as placebo.
  Interventions: Biological: recombinant HIV-1 Tat protein
- B (Other): Subjects were immunized intradermally with Tat, 3 dosage groups (7.5, 15 or 30 microgrammi), or with Saline, as placebo.
  Interventions: Biological: recombinant HIV-1 Tat protein

INTERVENTIONS:
Biological: recombinant HIV-1 Tat protein

SUMMARY:
The development of a vaccine against HIV/AIDS has been primary focused on the structural proteins (Env, Gag) of HIV-1 with the aim of inducing sterilizing immunity by blocking virus entry. Alternative approaches are focused on new vaccine strategies aimed at modifying the virus-host dynamic favouring the establishment of a long-term non-progressing disease status. Such strategies target regulatory proteins that are the first to be expressed after infection and are essential for viral replication, infectivity and pathogenesis. Thus, this approach may be effective for both preventive and therapeutic vaccination strategies.

DETAILED DESCRIPTION:
Being a very early viral regulatory protein necessary for viral gene expression, cell-to-cell virus transmission and disease progression, Tat represents a key target protein for the host immune response and an optimal candidate for such a vaccination strategy.

Preclinical studies demonstrated that vaccination with a biologically active Tat protein is safe, elicits a broad and specific immune response and induces a long-term protection against infection. Cross-sectional and longitudinal studies in natural infection suggest that the presence of an anti-Tat humoral immune response correlates with asymptomatic infection and with a slower disease progression while the presence of CD8+ T cell responses to Tat correlate with early virus control both in humans and monkeys. Since the immunogenic regions of Tat are well conserved among the HIV-1 M group, a vaccine based on Tat may be used in different geographic areas of the world.

This Phase I study was directed at evaluating the safety profile (as a primary end-point) and the immunogenicity (as a secondary end-point) of the recombinant HIV-1 Tat vaccine in HIV-1 infected adult volunteers with mild immune deficiency (Clinical category A according to CDC), CD4+ T cell counts 400/mL and levels of plasma viremia < 50,000 copies/mL.

Study Design: Randomized, Double Blind, Placebo Controlled, Safety/Immunogenicity Study.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test for women of childbearing potential within 3 days prior to baseline evaluation and use of an acceptable means of contraception (condom, hormonal or mechanical method) for one month prior to immunization and the duration of the study;
* Clinically asymptomatic HIV-1 infected individuals (CDC Clinical category A), as determined by two positive Enzyme-linked immunosorbent assay (ELISA) and a confirmatory Western Blot;
* Mean CD4+ T cell count >= 400 cells/microL based on 2 separate determinations, at least 2 weeks apart, within the four weeks pre-study screening period. [Note: If one of the two values is < 400 the patient will be excluded. Patients ever having had a value of CD4+ T cell number < 250 will be excluded];
* Plasma HIV-1 viremia levels <= 50,000 copies/mL;
* Complete blood count and differential defined as:
* Hematocrit >= 30% for women, >= 38% for men
* Hemoglobin >= 9.5 g/dL
* White cell counts >= 4,000 cells/mm3
* Total lymphocyte count >= 1000 cells/mm3
* Platelets >= 100,000/mm3
* Differential within institutional normal limits or approval of site physician
* Normal ALT (as defined by the range of the clinical site laboratories) and Creatinine (<= 1.6 mg/dL);
* Normal urine dipstick with esterase and nitrite;
* Normal thyroid function;
* Availability for follow-up for planned duration of at least 12 months and willing to have further brief evaluations at 24 and 36 months;
* Signed informed consent.

Exclusion Criteria:

* History of AIDS-related opportunistic or neoplastic disease;
* History of encephalopathy, neuropathy, or unstable CNS pathology (HIV or non-HIV related);
* History of non-HIV related neoplastic diseases, autoimmune diseases, angina or cardiac arthymias, or any other clinically significant medical problems;
* Chest radiography showing evidence of active or acute cardiac or pulmonary disease;
* History of anaphylaxis or serious adverse reactions to vaccines as well as serum IgE levels exceeding 1000 U.I./mL;
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g. Steven-Johnson syndrome, bronchospasm, or hypotension);
* Active syphilis [NOTE. If the serology is documented to be a false positive or due to an adequately treated infection, the volunteer is eligible];
* Active tuberculosis [NOTE: Volunteers with a positive PPD and a normal chest X-ray showing no evidence of TB and not requiring isoniazid (INH) therapy are eligible];
* Medical or psychiatric condition or occupational responsibilities which preclude subject compliance with the protocol. Specifically excluded are persons with psychotic disorders, major affective disorders, suicidal ideation;
* Current use of psychotrophic drugs;
* Use of antiretroviral therapy within 3 months of pre-study screening.
* Use of any experimental HIV therapy or participation in another experimental protocol within three (3) months of pre-study screening;
* Current or prior therapy with immunomodulators or immunosuppressive drugs and anticoagulant drugs within 30 days prior to study medication administration;
* Any unstable cardio-vascular disease (e.g unstable hypertensive disease needing modification or introduction of an anti-hypertensive treatment);
* Live attenuated vaccines within 60 days of study [NOTE: Medically indicated sub-unit or killed vaccines (e.g., influenza, pneumococcal, hepatitis A and B) are not exclusionary, but should be given at least 4 weeks away from HIV immunizations];
* Receipt of blood products or immunoglobulin in the past year;
* Prior receipt of HIV-1 vaccine in a previous HIV vaccine trial;
* Positivity for HBV antigens (HBs Ag, HBe Ag), and HCV, HTLV-I and HTLV-II antibodies;
* Positivity for HHV-8 antibodies and plasmaviremia (volunteers will be screened for anti-HHV-8 antibodies and positivity confirmed by PCR, only the individuals confirmed positive by PCR will be excluded);
* Pregnant or lactating women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2003-12; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Assessment of product safety included clinical monitoring of volunteers for local and systemic adverse reactions during the course of the trial and monitoring of haematological, biochemical, virological and immunological parameters

SECONDARY OUTCOMES:
To qualify Tat protein as immunogenic, volunteers were monitored for anti-Tat specific antibodies (IgM, IgG, IgA), anti-Tat proliferative response and in vitro γIFN and IL-4 production by PBMC before vaccination and in response to Tat vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ensoli, MD, PhD, Study Director — National AIDS Center, Istituto Superiore di Sanità, Rome, Italy
Locations (4):
- Italy (4):
  - San Raffaele Hospital, Milan
  - Hospital Spallanzani, Rome
  - San Gallicano Hospital, Rome
  - University of Rome "La Sapienza", Rome

REFERENCES:
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Cafaro A, Caputo A, Fracasso C, Maggiorella MT, Goletti D, Baroncelli S, Pace M, Sernicola L, Koanga-Mogtomo ML, Betti M, Borsetti A, Belli R, Akerblom L, Corrias F, Butto S, Heeney J, Verani P, Titti F, Ensoli B. Control of SHIV-89.6P-infection of cynomolgus monkeys by HIV-1 Tat protein vaccine. Nat Med. 1999 Jun;5(6):643-50. doi: 10.1038/9488. PMID 10371502
- [Background] Cafaro A, Caputo A, Maggiorella MT, Baroncelli S, Fracasso C, Pace M, Borsetti A, Sernicola L, Negri DR, Ten Haaft P, Betti M, Michelini Z, Macchia I, Fanales-Belasio E, Belli R, Corrias F, Butto S, Verani P, Titti F, Ensoli B. SHIV89.6P pathogenicity in cynomolgus monkeys and control of viral replication and disease onset by human immunodeficiency virus type 1 Tat vaccine. J Med Primatol. 2000 Aug;29(3-4):193-208. doi: 10.1034/j.1600-0684.2000.290313.x. PMID 11085582
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- See also: Related Info — http://www.iss.it